CLINICAL TRIAL: NCT02467010
Title: Bortezomib in Combination With Continuous Low-dose Oral Cyclophosphamide and Dexamethason Followed by Maintenance in Primary Refractory or Relapsed Bortezomib naïve Multiple Myeloma Patients. A Prospective Phase II Study.
Brief Title: Relapse Myeloma; Cyclofosfamide; Bortezomib; Maintenance
Acronym: REMM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, E. Vellenga, Prof.dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCG REMM; 2008-004822-17 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma
Keywords: Bortezomib; cyclophosphamide; dexamethason; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib, cyclophosphamide, dexamethason (Experimental): * To assess the efficacy of bortezomib, cyclophosphamide and dexamethasone during re-induction and in maintenance therapy.
  * To assess the safety of bortezomib, cyclophosphamide and dexamethasone during re-induction and in maintenance therapy in patients with refractory or relapsed multiple myeloma.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Re-induction chemotherapy with bortezomib, cyclophosphamide and dexamethasone. All patients with first relapse or primary refractory multiple myeloma and bortezomib naive will be given 6 cycles of re-induction therapy. Patients will be evaluated for response after cycle 3 and 6.
  Maintenance therapy with bortezomib and cyclophosphamide Maintenance therapy with bortezomib and cyclophosphamide will start at 4 weeks after the last cycle of re-induction chemotherapy if ANC ≥ 2.0 x 109/l and platelets > 75 x 109/l. Bortezomib is administered once every other week and cyclophosphamide (50 mg) every day for 1 year or until progression or death of any cause.
  Other Names: Velcade
Drug: Cyclophosphamide — Re-induction chemotherapy with bortezomib, cyclophosphamide and dexamethasone. All patients with first relapse or primary refractory multiple myeloma and bortezomib naive will be given 6 cycles of re-induction therapy. Patients will be evaluated for response after cycle 3 and 6.
  Maintenance therapy with bortezomib and cyclophosphamide Maintenance therapy with bortezomib and cyclophosphamide will start at 4 weeks after the last cycle of re-induction chemotherapy if ANC ≥ 2.0 x 109/l and platelets > 75 x 109/l. Bortezomib is administered once every other week and cyclophosphamide (50 mg) every day for 1 year or until progression or death of any cause.
  Other Names: Endoxan
Drug: Dexamethasone — Re-induction chemotherapy with bortezomib, cyclophosphamide and dexamethasone. All patients with first relapse or primary refractory multiple myeloma and bortezomib naive will be given 6 cycles of re-induction therapy. Patients will be evaluated for response after cycle 3 and 6.
  Maintenance therapy with bortezomib and cyclophosphamide Maintenance therapy with bortezomib and cyclophosphamide will start at 4 weeks after the last cycle of re-induction chemotherapy if ANC ≥ 2.0 x 109/l and platelets > 75 x 109/l. Bortezomib is administered once every other week and cyclophosphamide (50 mg) every day for 1 year or until progression or death of any cause.

SUMMARY:
Bortezomib and cyclophosphamide in combination with dexamethasone has already demonstrated high response rates in refractory multiple myeloma. Low dose continuous cyclophosphamide, also called metronomic scheduling, minimize toxic side effects and eliminate the obligatory rest periods. Combining cyclophosphamide with bortezomib might target distinct aspects of a myeloma functionality.

The objectives of the present study are whether patients with refractory or relapsed multiple myeloma after reinduction with bortezomib, cyclophosphamide and dexamethasone will benefit from maintenance therapy with bortezomib and cyclophosphamide with acceptable side-effects. Recently two studies have shown with thalidomide that maintenance therapy might improve EFS and one study also the OS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Stage II-III Multiple Myeloma
* Relapse or primary refractory disease after initial chemotherapy
* WHO performance status 0 - 2
* Life expectancy of at least 6 weeks
* ANC (absolute neutrophil count) ≥ 1.0x109/l(or ≥ 0.5x109/l, if due to bone marrow infiltration by malignancy)
* Platelet count ≥ 75x109/l or ≥ 50x109/l, if due to bone marrow infiltration by malignancy)
* Written informed consent (present in patient's file)
* Patient is able and willing to use adequate contraception during therapy and for at least 1 month after study
* Patient has the ability to understand the requirements of the study

Exclusion Criteria:

* Previous treatment with bortezomib
* Urine production < 1.5 l/24h
* Pre-existent polyneuropathy (grade 2 or higher, according to CTCAE 3.0)
* Pregnancy or positive pregnancy tests during study and for 1 month after final dose of thalidomide
* History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin)
* Active uncontrolled infections
* Additional uncontrolled serious medical or psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Toxicity of induction chemotherapy according to CTCAE version 3.0 | 5 years

SECONDARY OUTCOMES:
Progression Free Survival | 5 years
Overall Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sjoerd Hovenga, Principal Investigator — Nij Smellinghe Hospital Drachten
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands